CLINICAL TRIAL: NCT00309504
Title: Pulse Sequence Development on 3T Magnetic Resonance Imaging/Spectroscopy
Status: Completed | Type: Observational
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 22307
Record Dates: First submitted 2006-03-31; First posted 2006-04-03 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2012-03

CONDITIONS: Healthy
Keywords: magnetic resonance imaging; magnetic resonance spectroscopy

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to find ways to improve the appearance of tumours or markers that indicate the presence of tumours in Magnetic Resonance Imaging (MRI). Although based on the same technology, there are many ways to obtain images using MRI. The type of image that will be produced by the scanner depends on the instructions sent to the machine. These instructions tell different components of the machine when to turn on and off and all together are called a pulse sequence. These pulse sequences can get quite lengthy and intricate and small changes in them can produce considerable changes in the resulting image. the aim of this protocol is to alter existing pulse sequences to improve image appearance. This protocol will involve only healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult

Exclusion Criteria:

* subject under 18 years of age
* subject pregnant, or may be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Local Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2006-03; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gino B. Fallone, PhD, FCCPH, DABR, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada